CLINICAL TRIAL: NCT06913647
Title: Effect of Canagliflozin on Ultrafiltration and Fibrosis in Peritoneal Dialysis: a a Proof-of-concept Randomized Phase II Crossover Clinical Trial
Brief Title: Effect of Canagliflozin on Ultrafiltration & Fibrosis in Patients on Peritoneal Dialysis
Acronym: CAN-PD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Thomas Mavrakanas, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-11346
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: ESRD; CKD (Chronic Kidney Disease) Stage 5D
Keywords: SGLT-2 inhibitors; Canagliflozin; Ultrafiltration failure; Peritoneal fibrosis; Peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Peritoneal Fibrosis | interventions — Canagliflozin

STUDY DESIGN:
Intervention Model Description: This is a phase II, proof-of-concept, placebo-controlled, double-blind, cross-over randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The cross-over part of the study for the assessment of the primary outcome will be blinded (first 10 weeks for arms 1 & 2). Canagliflozin pills will be encapsulated. For placebo, cellulose will be used to fill identical capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active treatment followed by placebo (Active Comparator): Canagliflozin 300 mg once daily for 5 weeks (double-blind), followed by matching placebo once daily for 5 weeks (double-blind), followed by canagliflozin 300 mg once daily for 16 weeks (open label)
  Interventions: Drug: Canagliflozin 300 MG
- Placebo followed by active treatment (Placebo Comparator): Placebo once daily for 5 weeks (double-blind), followed by canagliflozin 300 mg once daily for 5 weeks (double-blind), followed by canagliflozin 300 mg once daily for 16 weeks (open label)
  Interventions: Drug: Canagliflozin 300 MG
- Standard of care (No Intervention): Standard of care, with no active treatment, for 26 weeks (open label)

INTERVENTIONS:
Drug: Canagliflozin 300 MG — Canagliflozin 300 mg once daily
  Other Names: Invokana 300 mg
  Arms: Active treatment followed by placebo; Placebo followed by active treatment

SUMMARY:
This is a phase II, proof-of-concept, placebo-controlled, double-blind, cross-over randomized clinical trial, assessing the effect of canagliflozin on peritoneal membrane function in patients on PD.

The primary aim of this trial is to determine the short-term effects of canagliflozin, an SGLT-2 inhibitor, on glucose absorption by the peritoneal membrane and on ultrafiltration, as assessed by a standardized peritoneal equilibrium test. The secondary aims are to determine the effect of canagliflozin on solute clearance and on effluent biomarkers of inflammation, angiogenesis, and fibrosis at 26 weeks. We hypothesize that canagliflozin will prevent glucose absorption by the peritoneal membrane, as compared with placebo, and will attenuate the development of inflammation, angiogenesis, and fibrosis of the peritoneal membrane, as assessed by relevant biomarkers in the dialysate.

DETAILED DESCRIPTION:
Patients with kidney failure on peritoneal dialysis who meet the study inclusion criteria will be randomized at a 2:2:1 ratio to one of the following arms:

(i) canagliflozin 300 mg once daily for 5 weeks (double-blind), followed by matching placebo once daily for 5 weeks (double-blind), followed by canagliflozin 300 mg once daily for 16 weeks (open label).

(ii) placebo once daily for 5 weeks (double-blind), followed by canagliflozin 300 mg once daily for 5 weeks (double-blind), followed by canagliflozin 300 mg once daily for 16 weeks (open label).

(iii) standard of care, with no active treatment, for 26 weeks (open label). Four in-person and one phone study visits have been scheduled: baseline visit, week 5, week 10, week 18 (phone visit), and week 26. A standardized peritoneal equilibration test (PET) will be performed at each of the in-person visits. There will also be two safety assessments at weeks 2 and 7, which will consist of blood tests. Patients who develop intercurrent illnesses or are hospitalized may temporarily discontinue the study drug if deemed appropriate by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with kidney failure on PD (both incident and prevalent) who are on a stable prescription of dextrose-based solutions for at least 3 months.
* Only high or high-average transporters, as classified by PET, will be included.

Exclusion Criteria:

* History of euglycemic ketoacidosis
* Known hypersensitivity to canagliflozin
* Active peritonitis or tunnel infection
* Kidney transplant scheduled in the next 6 months
* Severe liver cirrhosis (Child-Pugh class C stage)
* Recurrent severe genital or urine infections
* Patients receiving digoxin, phenobarbital, phenytoin, rifampin, or ritonavir if these agents cannot be safely discontinued
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in D4/D0 | 5 and 10 weeks from baseline
  Change in the ratio of intraperitoneal glucose at 0 and 4h post infusion (D4/D0 ratio) in a standardized PET with canagliflozin, compared with placebo.

SECONDARY OUTCOMES:
Change in ultrafiltration | 5 and10 weeks from baseline
  Change in ultrafiltration, as assessed by the volume of drain after a 4h dwell with 2 L of a 2.5% dextrose solution minus the volume infused, with canagliflozin compared with placebo.
Change in sodium dip/ sieving | 5 and 10 weeks from baseline
  Change in sodium dip/ sieving, calculated as the absolute difference in dialysate sodium at 0 and 1h post infusion in a standardized PET, with canagliflozin compared with placebo.
Change in small solute clearance | 5 and10 weeks from baseline
  Change in small solute clearance, as assessed by the dialysate-to-plasma (D/P) creatinine and urea at the end of a 4h-dwell, with canagliflozin compared with placebo.
Canagliflozin levels in the dialysate | 5 and10 weeks from baseline
  Canagliflozin levels in the dialysate at 5 and 10 weeks, as assessed by mass spectrometry
Change in small and middle solute clearance | 26 weeks from baseline
  Change in small and middle solute clearance using weekly Kt/V urea, weekly creatinine clearance, clearance of β2-microglobulin, and modifications in PD prescription.
Change in effluent biomarker levels | 26 weeks from baseline
  Change in effluent biomarker levels at 26 weeks from baseline. The panel of biomarkers includes interleukin-6 (IL-6), monocyte chemoattractant protein-1 (MCP-1), vascular endothelial growth factor (VEGF), cancer antigen-125 (CA-125), plasminogen activator inhibitor-1 (PAI-1), and decoy recptor-2 (eDcR2), assessed by using enzyme-linked colorimetric immunoassays.
Change in residual kidney function | 26 weeks from baseline
  Change in residual kidney function, as assessed by the 24h urine output and 24h native urea and creatinine clearance
Change in blood pressure | 26 weeks from baseline
  Change in 24h-ambulatory blood pressure measurements at 26 weeks from baseline
6-minute walk test | 26 weeks from baseline
  Change in distance in the 6-minute walk test at 26 weeks from baseline
Change in dyspnea score | 26 weeks from baseline
  Change in dyspnea score using the 7-point Likert scale and Visual analog scale questionnaire at 26 weeks from baseline
Change in quality of life | 26 weeks from baseline
  Difference in quality of life using the Kidney Disease Quality of Life questionnaire at 26 weeks from baseline
Major adverse cardiovascular events | 26 weeks from baseline
  Composite of cardiovascular death, myocardial infarction, stroke, hospitalization for heart failure
Death from any cause | 26 weeks from baseline
  Death from any cause
Safety outcomes | 26 weeks from baseline
  Safety outcomes, including serious adverse events and any adverse events

OTHER OUTCOMES:
Feasibility outcome | 26 weeks from baseline
  Ability to recruit for the study at the anticipated average recruitment rate and study completion with at least 80% adherence with reasons for non-adherence being reported

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Mavrakanas, MD, MSc., Principal Investigator — Research Institute-McGill University of Health Centre
Locations (1):
- Research Institute-McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
An anonymized dataset may be shared with other investigators in the future after the publication of primary results of this clinical trial. Any request for data sharing will have to be approved by the clinical trial steering committee after having examined the data sharing proposal. A data use agreement will be required through the Contracts Office of the Research Institute of McGill University Health Center.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data may become available twelve months after the end of the study.
Access Criteria: Any request for data sharing will have to be approved by the clinical trial steering committee after having examined the data sharing proposal. A data use agreement will be required through the Contracts Office of the Research Institute of McGill University Health Center.